CLINICAL TRIAL: NCT03242746
Title: The Effect of Cervical Morphological Changes on Pregnancy Outcome After Loop Electrosurgical Excision Procedure
Brief Title: Cervical Morphological Changes on Pregnancy Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-137
Record Dates: First submitted 2017-07-30; First posted 2017-08-08 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2017-09

CONDITIONS: Pregnancy Outcome
Keywords: LEEP; Loop Electrosurgical Excision Procedure; Cervical Intraepithelial Neoplasia; pregnancy outcome
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 1. The study will include 150 women of reproductive age (21-45 years) who wished to have future pregnancies and had cervical biopsy or Pap test, without any other cervical procedure, in the same calendar year.
  2. a 3-years follow-up for pregnancy outcome
  3. Transvaginal ultrasound for pretreatment cervical dimensions/volume
- LEEP group: 1. The study will include 150 women of reproductive age (21-45 years) planning for excisional treatment for CIN who wished to have future pregnancies. Women are included irrespective of their parity, previous obstetric history, and CIN grade.
  2. a 3-years follow-up for pregnancy outcome
  3. Transvaginal ultrasound for pretreatment cervical dimensions/volume
  4. Transvaginal ultrasound for posttreatment cervical dimensions/volume in the follow-up visit
  5. Estimation of cone dimensions/volume
  6. Calculation of the proportion of volume/length excised

SUMMARY:
This study aims to assess how the proportion of the cervical volume/length removed during treatment for cervical intraepithelial neoplasia (CIN) varies and whether this correlates to the pregnancy duration at delivery

DETAILED DESCRIPTION:
The high peak age of the Cervical intraepithelial neoplasia (CIN)patients was from 25 to 35 years old, which is the best women of childbearing age, Standard treatment for CIN is called Loop electrosurgical excision procedure (LEEP),but the inappropriate conization may damage the cervical function leading to infertility, abortion, preterm delivery and dystocia. Therefore, reasonable and standard conization is very important for treating and preventing the complication. The International Federation of Cervical Pathology and Colposcopy(IFCPC) advocates the length of cervical conization should be decided by the type of cervical transformation zone, however, the cervical lengths in female are different leading to the same cervical conization lengths cause the diverse influences on the cervical function.Therefore, individualized cervical conization therapies are very needed，At present, there are still lack of objective data about cervical morphology of women at childbearing age,besides the effects of cervical morphological changes caused by LEEP on pregnancy and childbirth has not been reported.

Our hypothesis is that the proportion of the cervical tissue removed is likely to influence both cervical healing and the cervical volume following surgery and as a result the risk of prematurity in subsequent pregnancies. The present prospective study investigates the variation in the proportion of the cervix removed during excisional treatment and provides pilot data on pregnancy outcomes in a sample population for which the dimensions and proportions of the cervical tissue excised are assessed at the time of treatment.

ELIGIBILITY:
Inclusion Criteria:

Having fertility requirements,antecedent biopsy read as

1. cervical intraepithelial neoplasia (CIN) grade 2 or 3 or microinvasive cancer
2. adenocarcinoma in situ
3. persistent CIN 1
4. antecedent pap read as
5. high grade squamous intraepithelial lesion
6. atypical glandular cells
7. persistent low grade squamous intraepithelial lesion

Exclusion Criteria:

1. anatomy unsuitable for safe office loop excision based on operator judgement
2. inability to tolerate procedure under local anesthesia
3. pregnancy
4. age less than 21 years
5. refusal of consent
6. prisoner
7. mental incapacity
8. anticoagulant or antiplatelet therapy, or known bleeding diathesis
9. use of analgesics other than over the counter medications(OTC meds include NSAIDS or Tylenol) within 7 days of scheduled LEEP.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Study Population: Women (18-45 y) plan for excisional CIN treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
pretreatment cervical dimensions/volume | at 24months
  The dimensions and volume of the cervix before treatment are calculated by two-dimensional transvaginal sonography (2D-TVS)
cone dimensions/volume | at 24months
  The dimensions of the cone are measured with a measuring tape and a ruler before formalin fixation. The measurements included the length/depth, and the anteroposterior,transverse, and lateral diameters. A fluid filled volumetric cylindrical vial (tube) are subsequently used to measure the cone volume with the fluid displacement technique
posttreatment cervical dimensions/volume | up to 12months
  Assessment of the cervical dimensions and the cervical volume is repeated 1,3,6,12 months post-treatment follow-up visit, using the same imaging technique as that used pretreatment
Pregnancy outcome | up to 48 months
  In the event of a pregnancy, the prenatal management and outcomes are recorded. More specifically, it is recorded whether interventions such as cervical length ultrasound, cervical cerclage, or progesterone are used. The duration of pregnancy at delivery, the birth weight, and other obstetric outcomes and complications are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Hu, Study Chair — The Second Affiliated Hospital of Chongqing Medical University; Shufang Chang, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Hu Li, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- 2ndChongqingMU, Yuzhong, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalliala I, Anttila A, Nieminen P, Halttunen M, Dyba T. Pregnancy incidence and outcome before and after cervical intraepithelial neoplasia: a retrospective cohort study. Cancer Med. 2014 Dec;3(6):1512-6. doi: 10.1002/cam4.300. Epub 2014 Aug 21. PMID 25146172
- [Background] Kalliala I, Anttila A, Dyba T, Hakulinen T, Halttunen M, Nieminen P. Pregnancy incidence and outcome among patients with cervical intraepithelial neoplasia: a retrospective cohort study. BJOG. 2012 Jan;119(2):227-35. doi: 10.1111/j.1471-0528.2011.03042.x. Epub 2011 Jul 27. PMID 21790950